CLINICAL TRIAL: NCT05184725
Title: CARINAE: A Digital Health Intervention for Stress Relief in Perioperative Care: Clinical Study
Brief Title: CARINAE for Stress Relief in Perioperative Care
Acronym: CARINAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adhera Health, Inc. (Industry)
Collaborators: Maastricht University Medical Center (Other); Hospital Sant Joan de Deu (Other); Parc Taulí Hospital Universitari (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government); Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAR-0320
Record Dates: First submitted 2021-11-29; First posted 2022-01-11 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Psychological Stress; Cardiopulmonary Bypass Surgery; Coronary Artery Bypass Surgery; Cardiac Valve Replacement; Hip Replacement; Orthognathic Surgery; Scoliosis; Knee Replacement; Prostate Cancer; Kidney Cancer; Bladder Cancer
Keywords: Pre-operative Stress; mHealth Device; Virtual Reality (VR); Health Recommender System; I-Change Behavioral Change Model; Artificial Intelligence (AI); Software as a Medical Device (SaMD)
MeSH Terms: conditions — Stress, Psychological; Scoliosis; Prostatic Neoplasms; Kidney Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: The SaMD CARINAE embeds the I-Change Model, which claims that behavioral changes depend on the inner motivation to perform a specific behavior and the self-perception of personal abilities, or self-efficacy perception, to carry out the behavioral change.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients will follow the usual care procedures and after each procedure they answer questionnaires related to pain and stress levels (VAS), Anxiety and depression levels (HADS), health-related quality of life (HRQoL), mental wellbeing (SWEMWBS), self-efficacy (GSE) and Patient Activation status (PAM-13).
- SaMD CARINAE (Experimental): Intervention group will be exposed to the use of SaMD CARINAE for 2 months approximately, a patientcentred digital health support program. The intervention trial will include a total of 4 visits: 1. Baseline (2-4 weeks before surgery); 2. Hospital admission (1-3 days before surgery); 3. Hospital discharge (1 week after the surgery approx.); 4. Post-operative day 14 (2 weeks after the surgery approx). After each visit and intervention trial with SaMD CARINAE the experimental group answer the same questionnaires of the control group, above mentioned Participants allocated to the intervention group will also be asked to complete questionnaires about usability, satisfaction and subjective experience.
  Interventions: Device: SaMD CARINAE

INTERVENTIONS:
Device: SaMD CARINAE — SaMD CARINAE delivers the following digital therapeutic intervention to the patients: 1) Personalised patient-centred health education program to improve patient's disease and recovery self-management skills. 2) AI-based behaviour change program to promote healthier lifestyle habits. 3) Personalised mental well-being coaching program to improve patient's ability to cope with emotional disturbances such as stress and anxiety. 4) A collaborative digital support platform to enable information exchange between patients, caregivers, and healthcare professionals.
  Arms: SaMD CARINAE

SUMMARY:
Preventing pre-surgical stress can help patients achieve positive outcomes on health and well-being. However, very few patients receive adequate stress relief support prior to a surgical procedure. Provision of education and information about the surgery can be a crucial component of the preoperative experience and is inversely related to levels of preoperative anxiety. However, resource constraints make face-to-face education sessions untenable, given cost considerations and time investment by trained health personnel. Interventions based on mobile health (mHealth) technologies, geared towards increasing familiarity with surgical procedures and hospital environments have been shown to help patients feel informed about possible benefits and risks of available treatment options. mHealth apps and Virtual Reality (VR) can offer patients experience in the perioperative environment that can be helpful in empowering patients and enhancing a more positive experience, while reducing stress. However, available applications focus only on providing informative content, neglecting the importance of patient empowerment with a more robust educational curriculum.

According to this, the Software as a Medical Device (SaMD) CARINAE, aims to support patients and caregivers during the whole perioperative process. SaMD CARINAE consists of an mHealth mobile application for patients and caregivers, a Virtual Reality headset for patients, and a web application for healthcare professionals.

DETAILED DESCRIPTION:
Patients will be randomly assigned to intervention group or the control group. Intervention group will be exposed to the use of SaMD CARINAE for 2 months approximately. The intervention trial will include a total of 4 visits: 1. Recruitment; 2. Hospital admission; 3. Hospital discharge; 4. Post-operative follow-up in 14 days.

SaMD CARINAE delivers the following interventions to the patients:

* Personalised patient-centred health education program to improve patient's condition and recovery self-management skills.
* Artificial Intelligence-based behaviour change program to promote healthier lifestyle habits.
* Personalised mental well-being coaching program to improve patient's ability to cope with emotional disturbances such as stress and anxiety.
* A collaborative digital support platform to enable information exchange between patients, caregivers, and healthcare professionals.

The program is delivered to patients and caregivers as a SaMD mHealth application (smartphone app) and an immersive environment with a VR device. Healthcare professionals will be able to access the collaborative digital support platform through a web application.

Finally, the control group will not be exposed to SaMD CARINAE solution, following the traditional routine visits, and after each traditional visit patients will answer to questionnaires specified in the secondary outcome measures section.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for one of the selected surgery types:
* Cardiopulmonary bypass (CPB) surgery (Maastricht UMC+)
* Coronary artery bypass surgery (Maastricht UMC+)
* Cardiac valve replacement (SAS, Maastricht UMC+)
* Prostate, kidney, and bladder cancer surgery (INRCA)
* Hip and knee replacement (HSJD; Parc Tauli)
* Maxillofacial surgery (HSJD)
* Orthognathic surgery (HSJD)
* Scoliosis (HSJD)
* Signed informed consent (by patient or legal guardian in paediatric cases).
* Patients ≥ 18 years old, except for paediatric Hospital San Joan de Deu (HSJD) ≥ 8 years old.
* Patient owns a smartphone with Android version 4.4 or above.
* Patient (or legal guardian/caregiver in paediatric cases) is able to demonstrate basic digital literacy (e.g. knows how to communicate through instant messaging apps or similar).

Exclusion Criteria:

* Dementia.
* Pregnant women.
* Inability to understand the local language.
* Allergic to dedicated wearable material (stainless steel and silicone).
* Currently enrolled in a different clinical trial.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for Stress | 2 months: from baseline to 14 days after the surgery
  Patient and caregiver-reported visual analog scale question to assess subjective stress.
  Along a 100 mm horizontal line, patient and caregiver indicate their perceived stress intensity. Rating varies from 0 (minimum values) to 100 (maximum value). Ratings of 0 to 4 mm can be considered no stress; 5 to 44 mm, mild stress; 45 to 74 mm, moderate stress; and 75 to 100 mm, severe stress.
Visual Analog Scale for Pain | 2 months: from baseline to 14 days after the surgery
  Patient-reported visual analog scale question to assess subjective pain. Along a 100 mm horizontal line, patient and caregiver indicate their perceived pain intensity. Rating varies from 0 (minimum values) to 100 (maximum value). Ratings of 0 to 4 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain.
Hospital Anxiety and Depression Scale | 45 days: From hospital admission to 14 days after the surgery
  Patient-reported questionnaire on anxiety and depression levels during the hospital stay. Hospital Anxiety and Depression Scale is a fourteen-item scale with seven items each for anxiety and depression subscales evaluated on a 0-3 Likert Scale. Rating varies from 0 to 21 and a subscale score >8 denotes anxiety or depression.
Health-related Quality of Life - EQ-5D-3L/-Y | 45 days: From hospital admission to 14 days after the surgery
  Patient-reported questionnaire on quality of life. The questionnaire consists of five items related each to one dimension: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems (1), some problems (2), and extreme problems (3). The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status with 100 indicating the best health status.
The Positive and Negative Affect Schedule | 45 days: From hospital admission to 14 days after the surgery
  Patient-reported questionnaire on emotional status. It consists of 20 items that describe n emotions of a positive or negative nature, 10 of them positive and 10 negative. Each item is answered using an Likert-tscale with 5 response options (not at all, very little, somewhat, quite a lot, very much).
  Scores can range from 10 - 50, with higher scores representing higher levels of positive or negative affect.
The Short Warwick-Edinburgh Mental Well-Being Scale | 2 months: from baseline to 14 days after the surgery
  Patient- and caregiver-reported questionnaire on mental well-being. It consists of 7 items and each item is answered using a 1-5 Likert scale. Scores range from 7 to 35 and higher scores indicate higher positive mental wellbeing.
General Self-Efficacy Scale | 2 months: from baseline to 14 days after the surgery
  Patient- and caregiver-reported questionnaire on self-efficacy perception. It consists of 10 items evaluated on a 1-4 Likert scale. Scores range from 10 to 40 amd higher scores indicate higher self-efficacy.
Patient Activation Measure | 45 days: From baseline to hospital discharge
  Patient-reported questionnaire on the level of activation. It consists of 13 items that have four possible response options ranging from (1) strongly disagree to (4) strongly agree, and an additional "not applicable" option. To calculate the total score, the raw score is divided by the number of items answered (excepting non-applicable items) and multiplied by 13. Then, this score is transformed to a scale with a theoretical range 0-100, based on calibration tables, with higher scores indicating higher patient activation. The raw scores can be converted into four activation levels: 1 (≤47.0) not believing activation important, 2 (47.1-55.1) a lack of knowledge and confidence to take action, 3 (55.2-67.0) beginning to take action and 4 (≥67.1) taking action.

SECONDARY OUTCOMES:
System Usability Scale | 30 days: from hospital admission to 14 days after surgery
  Questionnaire on SaMD CARINAE usability by patients, caregivers and healthcare professionals
Usability questionnaire | 30 days: from hospital admission to 14 days after surgery
  Ad-hoc questionnaire for patients and healthcare professional on the digital solution usability
Net Promoter Score | 30 days: from hospital admission to 14 days after surgery
  Net Promoter Score (NPS) is a questionnaire that measures patient and healthcare professionals experience and provides the core measurement for customer experience management programs.
Reliability | Day 60
  Ad-Hoc questionnaire for the healthcare professional on the digital solution

CONTACTS AND LOCATIONS:
Overall Officials: Clara Hernández Cera, Principal Investigator — Hospital San Joan de Deu; Ignacio Muñoz Carvajal, Study Director — Hospital Universitario Reina Sofía; Juan José Lázaro Alcay, Study Chair — Hospital San Joan de Deu; Andrea Vallejo Tarrat, Study Chair — Parc Taulí Hospital Universitari; JG Maessen, Prof. dr., Study Chair — Maastricht University Medical Center; Marco Dellabella, Study Chair — Istituto di Ricovero e Cura per Anziani
Locations (5):
- Istituto di Ricovero e Cura per Anziani, Ancona, Italy
- Maastricht University Medical Center, Maastricht, Netherlands
- Spain (3):
  - Hospital Reina Sofía, Córdoba, Andalusia
  - Hospital San Joan de Deu, Esplugues de Llobregat, Catalonia
  - Hospital Parc Taulí, Sabadell, Catalonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crichton, N. Visual analogue scale (VAS). J Clin Nurs. 2001; 10(5): 706-6.
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398
- [Background] Schwarzer, R., & Jerusalem, M. Generalized Self-Efficacy scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs. Windsor, UK: NFER-NELSON. 1995; 35-37.
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Brooke, J. SUS-A quick and dirty usability scale. Usability evaluation in industry. 1996; 189(194): 4-7.
- [Background] Reichheld FF. The one number you need to grow. Harv Bus Rev. 2003 Dec;81(12):46-54, 124. PMID 14712543
- [Derived] Kondylakis H, Giglioli IAC, Katehakis D, Aldemir H, Zikas P, Papagiannakis G, Hors-Fraile S, Gonzalez-Sanz PL, Apostolakis K, Stephanidis C, Nunez-Benjumea FJ, Banos-Rivera RM, Fernandez-Luque L, Kouroubali A. Stress Reduction in Perioperative Care: Feasibility Randomized Controlled Trial. J Med Internet Res. 2025 Jan 7;27:e54049. doi: 10.2196/54049. PMID 39773866
- [Derived] Kondylakis H, Chicchi Giglioli IA, Katehakis DG, Aldemir H, Zikas P, Papagiannakis G, Hors-Fraile S, Gonzalez-Sanz PL, Apostolakis KC, Stephanidis C, Nunez-Benjumea FJ, Banos-Rivera RM, Fernandez-Luque L, Kouroubali A. A Digital Health Intervention for Stress and Anxiety Relief in Perioperative Care: Protocol for a Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2022 Nov 29;11(11):e38536. doi: 10.2196/38536. PMID 36445734